CLINICAL TRIAL: NCT06366880
Title: Parenteral Nutrition Cycling for Prevention of Cholestatic Syndrome in Newborn
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Pediátrico de Sinaloa (Other Government)
Responsible Party: Principal Investigator, Camargo Angulo Ana Karen, Dr., Hospital Pediátrico de Sinaloa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2022.HPS.DI.434
Record Dates: First submitted 2024-03-11; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Cholestasis in Newborn
Keywords: Parenteral nutrition cycling; Incidence of colestasis; Incidence of hypoglycemia; Hospital-acquired infections; Randomised controlled trial

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parenteral nutrition cycling (Experimental)
  Interventions: Other: Parenteral nutrition cycling
- Continuous parenteral nutrition (No Intervention)

INTERVENTIONS:
Other: Parenteral nutrition cycling — This study is a single-centre, non-blinded RCT in the NICU of Pediatric Hospital of Sinaloa, Northwest, Mexico.
  A total of 66 infants born ≥34 weeks of gestation who have a high likelihood of intolerance to enteral nutrition (EN) for at least 10 days will be randomised to PNC o PNT after informed parental consent. In both groups, EN will be commenced as early as clinically feasible.
  Other Names: Cyclic parenteral nutrition; Cycling parenteral nutrition; Cycle parenteral nutrition
  Arms: Parenteral nutrition cycling

SUMMARY:
Background: Despite the use of parenteral nutrition cycling (PNC) in neonatal intensive care units (NICU), there is limited evidence regarding the benefits in relation to the nutrición parenteral total (NPT) in term and late preterm infants.

The recommendations from the recently published Latin American Society of Gastroenterology, Hepatology and Pediatric Nutrition guidelines are substantially different in this area, and surveys have reported variations in clinical practice.

The aim of this randomised controlled trial (RCT) is to evaluate the benefits and risks of PNC AND parenteral nutrition total (NPT) in term and late preterm infants.

DETAILED DESCRIPTION:
Methods/design:

This study is a single-centre, non-blinded RCT in the NICU of Pediatric Hospital of Sinaloa, Northwest, Mexico.

A total of 66 infants born ≥34 weeks of gestation who have a high likelihood of intolerance to enteral nutrition (EN) for at least 10 days will be randomised to PNC o PNT after informed parental consent. In both groups, EN will be commenced as early as clinically feasible.

Primary outcomes Incidence of colestasis on Day 28 of admission.

Secondary outcomes are total plasma bilirrubine profiles, the incidence of hypoglycemia, hospital-acquired infections, length of hospital/NICU stay, in-hospital all-cause mortality, weight, height and head circumference.

Discussion: This RCT will examine the effects of NPTC versus late PNT in term and late preterm infants by comparing key biochemical and clinical outcomes and has the potential to identify underlying pathways for beneficial or harmful effects related to both treatments.

Trial registration: 2022.HPS.DI.434 (3rd March 2024)

Keywords: Parenteral nutrition cycling, Incidence of colestasis, incidence of hypoglycaemia, hospital-acquired infections, Randomised controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Chylothorax
* Intestinal obstruction
* Intestinal malrotation
* Intestinal intussusception
* Gastroschisis
* Intestinal volvulus
* Duodenal atresia
* Enterocolitis
* Sepsis
* Septic shock
* Prolonged fast
* Authorization of the study by parents

Exclusion Criteria:

* Presence of liver diseases or malformations that cause cholestasis.
* All patients who have received medical treatment for cholestasis are excluded.

Ages: 1 Hour to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2024-12-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of cholestasis on Day 28 of admission. | Day 1 to 28
  Proportion of cholestasis

SECONDARY OUTCOMES:
are total plasma bilirrubine profiles | Day 1 to 28
  mg/dl
the incidence of hypoglycaemia | Day 1 to 28
  mg/dl

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Pediatrico de Sinaloa, Culiacán, Sinaloa, Mexico